CLINICAL TRIAL: NCT05787756
Title: Constipation and Changes in the Gut Flora in Parkinson's Disease: a Pilot Study
Brief Title: Constipation and Changes in the Gut Flora in Parkinson's Disease
Acronym: GUT-PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: Biomathematics & Statistics Scotland (BioSS) (Unknown); NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-048-21
Record Dates: First submitted 2023-03-01; First posted 2023-03-28 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — two stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson disease: Participants with newly diagnosed Parkinson's disease
- Control Subjects: Control subjects - will be selected from household/spousal contacts of the participants with Parkinson's disease

SUMMARY:
The aim of this study is to investigate the link between gut health and Parkinson's disease

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common, age-related neurological condition, affecting approximately 145,000 people in the United Kingdom. Diagnostic symptoms include stiffness, tremor, unsteadiness and slow movements. Interestingly, while PD is usually considered to be a neurological condition, pathological changes occur in the gut years before diagnosis, often causing constipation. As such, the gut has attracted attention as a possible therapeutic target.

Previous studies have shown different profiles of gut bacteria and the short chain fatty acids (SCFAs) they produce in people with PD. There is evidence these changes might be significant to the disease course, as faecal transplants from people with PD worsened symptoms in a mouse model of PD. The mechanism for this is unclear, but changes in SCFAs and gut wall inflammation, have both been suggested. Studies so far have compared gut bacteria in people with and without PD, however, as the healthy controls often don't have constipation, it is unclear if the differences seen are due to PD itself or the associated constipation.

This pilot study aims to determine differences in the frequency of gut micro-organisms (bacteria, fungi and archaea) and gut function, other than those caused by constipation. 40 participants with a new diagnosis of PD will be recruited from Movement Disorder clinics within National Health Service (NHS) Grampian. 40 healthy (non-PD) controls will be recruited from the PD participants households (whenever feasible). All 80 participants will be clinically assessed and asked to provide two stool samples. The samples will be analysed for the frequency of gut micro-organisms, changes in gut function (short chain fatty acid concentrations) and gut inflammation (calprotectin concentrations).

The aim of this pilot study is to determine the key differences in gut micro-organisms in PD compared to controls, which may have a role in disease progression. It is likely that the results of this proof of concept study would need to be confirmed in a larger study before the investigators are able to plan an intervention trial, such as testing a prebiotic product, with the aim of normalising gut micro-organisms, and potentially modifying the disease course.

ELIGIBILITY:
Inclusion Criteria:

Participants with Parkinson's disease 2. Community-dwelling patients with newly diagnosed PD who have not yet started medication for Parkinson's disease.

Control Participants

1. Healthy (non-Parkinsonian) members of the participants household will be invited to act as controls.

Exclusion Criteria:

1. Use of oral or intravenous antibiotics in the last 8 weeks.
2. Active gastrointestinal disease, not including constipation or irritable bowel syndrome without other symptoms.
3. Current use of medications which cause/worsen constipation e.g., opioids, tramadol, gabapentin, pregabalin.
4. Potential controls will be excluded if they report prodromal symptoms of PD, such as anosmia or rapid eye movement (REM) sleep disorder or display parkinsonian signs on examination.
5. Inability to give informed consent at any stage of the study e.g., because of dementia.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson disease group: potential participants will be invited into the study if they have recently been diagnosed with Parkinson's disease and have not yet started medication for the condition
  Control group: spouses or other household contacts will be invited to the study
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Micro-organism prevalence in stool sample | Baseline
  Stool samples will be posted to the Rowett Institute, and processed and analysed in the laboratory at The Rowett Institute, University of Aberdeen. The samples will be analysed for water content and microbial RNA/DNA will be extracted for genome analysis. When the analysis is complete, the faecal samples will be destroyed.
Micro-organism prevalence in stool sample | Within two months of baseline
  Stool samples will be posted to the Rowett Institute, and processed and analysed in the laboratory at The Rowett Institute, University of Aberdeen. The samples will be analysed for water content and microbial RNA/DNA will be extracted for genome analysis. When the analysis is complete, the faecal samples will be destroyed.

SECONDARY OUTCOMES:
Analysis of stool samples for concentration of short chain fatty acids | Baseline
  Stool samples will be posted to the Rowett Institute via Royal Mail. Samples will be processed and analysed in the laboratory at The Rowett Institute, University of Aberdeen. The samples will be analysed for short chain fatty acid concentration (µmol/g).
Analysis of stool samples for concentration of calprotectin | Baseline
  Stool samples will be posted to the Rowett Institute via Royal Mail. Samples will be processed and analysed in the laboratory at The Rowett Institute, University of Aberdeen. The samples will be analysed for short calprotectin concentration (µg/g).
Analysis of stool samples for markers of gut function (short chain fatty acids and calprotectin) | Within two months of the baseline sample
  Stool samples will be posted to the Rowett Institute via Royal Mail. Samples will be processed and analysed in the laboratory at The Rowett Institute, University of Aberdeen. The samples will be analysed for short chain fatty acid (SCFA) profile and calprotectin concentration. When the analysis is complete, the faecal samples will be destroyed.
To assess the extent of swallowing problems (dysphagia) by a questionnaire | Baseline
  Participants will be asked to completed a standardized swallowing questionnaire (Swallowing Disturbance Questionnaire), which has been validated in people with Parkinson's disease. The score ranges from 0-43, with a higher score increasing the likelihood for a swallowing problem, which would require further investigation
To assess the extent of swallowing problems using a standardized swallowing test | Baseline
  Participants will be asked to drink 150 millilitres of cold water from a clear cup. The rater will sit at their side and record them on video for later analysis. The speed in ml/second and volume per average swallow will be recorded by determining if any residual volume is left, the number of seconds to complete the task and the number of swallows. The test will be terminated if there is any indication of aspiration of liquid.
To assess the extent of swallowing problems using a standardized swallowing test | Four weeks after the baseline assessment
  Participants will be asked to drink 150 millilitres of cold water from a clear cup. The rater will sit at their side and record them on video for later analysis. The speed in ml/second and volume per average swallow will be recorded by determining if any residual volume is left, the number of seconds to complete the task and the number of swallows. The test will be terminated if there is any indication of aspiration of liquid.
To assess taste sensation using a simple test | Baseline
  Participants taste recognition will be assessed using standardized taste strips from Burghart (sweet, salty, sour and bitter)
To assess dietary intake over a 24 hour period using a structured interview | Baseline
  Following the initial visit, the participant will receive a phone call from a trained member of the team to perform a 24-hour dietary recall interview. This is a structured interview where participants are asked to recall all food and beverage consumption over a 24-hour period and further questions are asked to determine further details, including portion size and ingredients and cooking methods used. The whole interview usually takes 20 to 60 minutes.
To assess the reliability of bio-impedence analysis in determining fat mass in older adults with and without PD | Baseline
  Fat mass in kilograms will be measured using a seca mBCA 525 bio-impedence machine.
To assess the reliability of bio-impedence analysis in determining fat mass in older adults | Four weeks after baseline assessment
  Fat mass in kilograms will be measured using a seca mBCA 525 bio-impedence machine.
To assess the reliability of bio-impedence analysis in determining fat mass in older adults | Baseline
  Fat free mass in kilograms will be measured using a seca mBCA 525 bio-impedence machine.
To assess the reliability of bio-impedence analysis in determining fat mass in older adults | Four weeks after the baseline assessment
  Fat free mass in kilograms will be measured using a seca mBCA 525 bio-impedence machine.

CONTACTS AND LOCATIONS:
Overall Officials: Isobel JM Sleeman, BMBCh, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Human Nutrition Unit, Rowett Institute, University of Aberdeen, Aberdeen, Aberdeen City, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gage H, Kaye J, Kimber A, Storey L, Egan M, Qiao Y, Trend P. Correlates of constipation in people with Parkinson's. Parkinsonism Relat Disord. 2011 Feb;17(2):106-11. doi: 10.1016/j.parkreldis.2010.11.003. Epub 2010 Dec 3. PMID 21130017
- [Background] De Pablo-Fernandez E, Gebeyehu GG, Flain L, Slater R, Frau A, Ijaz UZ, Warner T, Probert C. The faecal metabolome and mycobiome in Parkinson's disease. Parkinsonism Relat Disord. 2022 Feb;95:65-69. doi: 10.1016/j.parkreldis.2022.01.005. Epub 2022 Jan 13. PMID 35045378
- [Background] Hilton D, Stephens M, Kirk L, Edwards P, Potter R, Zajicek J, Broughton E, Hagan H, Carroll C. Accumulation of alpha-synuclein in the bowel of patients in the pre-clinical phase of Parkinson's disease. Acta Neuropathol. 2014 Feb;127(2):235-41. doi: 10.1007/s00401-013-1214-6. Epub 2013 Nov 17. PMID 24240814
- [Background] Jaffrin MY, Morel H. Body fluid volumes measurements by impedance: A review of bioimpedance spectroscopy (BIS) and bioimpedance analysis (BIA) methods. Med Eng Phys. 2008 Dec;30(10):1257-69. doi: 10.1016/j.medengphy.2008.06.009. Epub 2008 Aug 3. PMID 18676172
- [Background] Manor Y, Giladi N, Cohen A, Fliss DM, Cohen JT. Validation of a swallowing disturbance questionnaire for detecting dysphagia in patients with Parkinson's disease. Mov Disord. 2007 Oct 15;22(13):1917-21. doi: 10.1002/mds.21625. PMID 17588237
- [Background] Mueller C, Kallert S, Renner B, Stiassny K, Temmel AF, Hummel T, Kobal G. Quantitative assessment of gustatory function in a clinical context using impregnated "taste strips". Rhinology. 2003 Mar;41(1):2-6. PMID 12677732
- [Background] Sampson TR, Debelius JW, Thron T, Janssen S, Shastri GG, Ilhan ZE, Challis C, Schretter CE, Rocha S, Gradinaru V, Chesselet MF, Keshavarzian A, Shannon KM, Krajmalnik-Brown R, Wittung-Stafshede P, Knight R, Mazmanian SK. Gut Microbiota Regulate Motor Deficits and Neuroinflammation in a Model of Parkinson's Disease. Cell. 2016 Dec 1;167(6):1469-1480.e12. doi: 10.1016/j.cell.2016.11.018. PMID 27912057
- [Background] Schwiertz A, Spiegel J, Dillmann U, Grundmann D, Burmann J, Fassbender K, Schafer KH, Unger MM. Fecal markers of intestinal inflammation and intestinal permeability are elevated in Parkinson's disease. Parkinsonism Relat Disord. 2018 May;50:104-107. doi: 10.1016/j.parkreldis.2018.02.022. Epub 2018 Feb 12. PMID 29454662
- [Background] Unger MM, Spiegel J, Dillmann KU, Grundmann D, Philippeit H, Burmann J, Fassbender K, Schwiertz A, Schafer KH. Short chain fatty acids and gut microbiota differ between patients with Parkinson's disease and age-matched controls. Parkinsonism Relat Disord. 2016 Nov;32:66-72. doi: 10.1016/j.parkreldis.2016.08.019. Epub 2016 Aug 26. PMID 27591074